CLINICAL TRIAL: NCT03864276
Title: The Comparison of Changes of QTc, Tp-e Interval, and Tp-e/QT Ratio, Tp-e/QTc Ratio on the ECG During Living Donor Liver Transplantation Under Desflurane and Total Intravenous Anesthesia -Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 4-2018-1164
Record Dates: First submitted 2019-03-04; First posted 2019-03-06 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Liver Cirrhosis(Who Will Undergo Planed Liver Transplantation)
MeSH Terms: interventions — Inhalation; Desflurane; Population Groups; Propofol; Anesthesia

STUDY DESIGN:
Intervention Model Description: Arm 1: inhalation anesthesia (desflurane) group Arm 2: total intravenous anesthesia (propofol) group
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: patients will be randomly allocated to 2 groups using computer-generated randomization method. Care provider will not be blinded to the group allocation, because anesthesiologists should be aware of the method of anesthesia.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- inhalation anesthesia (desflurane) group (Experimental): Anesthesia is induced and maintained with desflurane and sufentanil
  Interventions: Drug: inhalation (desflurane) group
- Total intravenous anesthesia (propofol) group (Experimental): Anesthesia is induced and maintained with propofol and sufentanil
  Interventions: Drug: total intravenous (propofol) anesthesia

INTERVENTIONS:
Drug: inhalation (desflurane) group — Anesthesia is induced and maintained with desflurane and sufentanil
  Arms: inhalation anesthesia (desflurane) group
Drug: total intravenous (propofol) anesthesia — Anesthesia is induced and maintained with propofol and sufentanil
  Arms: Total intravenous anesthesia (propofol) group

SUMMARY:
Prolonged corrected QT interval (QTc) has been observed in about half of patients with liver cirrhosis. Marked prolongation of QTc (ie, 500 msec) has been considered to be a risk factor for fatal ventricular arrhythmia, such as torsade de pointes,7,8 which has been reported in liver transplantation (LT) surgery. In a previous study, prolonged QTc interval ( 500 msec) was frequently observed throughout the procedure of LT, even among patients with baseline QTc 440 msec. Therefore, it is important to optimize electrolyte balance and hemodynamic status to reduce greater risk of perioperative arrhythmias.

The investigators hypothesized that the change of QTc interval might be differ according to method of general anesthesia (inhalation agent vs. intravenous agent).

ELIGIBILITY:
Inclusion Criteria:

* patients with liver cirrhosis who will undergo planned liver transplantation

Exclusion Criteria:

* 1. emergent liver transplantation
* 2. unstable angina
* 3. recent MI(Myocardial Infarction)
* 4. uncontrolled hypertension (diastolic BP > 110mmHg)
* 5. implantable cardiac defibrillator
* 6. severe obesity (BMI>30kg/m2)
* 7. allergy to propofol

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-02-17 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
QTc interval | 3 minutes after liver reperfusion
  The investigator will assess the QTc interval 3 minutes after the reperfusion during liver transplantation.

SECONDARY OUTCOMES:
QTc interval | at the end of the surgery
  The investigator will assess the QTc interval at the end of liver transplantation.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: Data will become available when the script for this study is accepted in journal.